CLINICAL TRIAL: NCT04622410
Title: Registry for Hirschsprung Disease of the BELAPS (Belgian Association of Pediatric Surgery)
Brief Title: Registry for Hirschsprung Disease of the BELAPS
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S51836
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Registry for Hirschsprung disease of the BELAPS (Belgian Association of Pediatric Surgery) Protocol Short Title/Acronym

/ Sponsor name BELAPS Principal Investigator Prof. Dr. Marc Miserez Medical condition or disease under investigation Hirschsprung's disease Purpose of clinical study To register pre-, intra- and postoperative data in order to improve surgical care to paediatric patients with Hirschsprung's disease in Belgium. Primary objective The primary objective is to evaluate defecation habits at 3.5-5.5 years after surgery. Secondary objective (s) Evaluating the long-term results and evaluate risk factors for constipation / incontinence. Study Design Prospective registry Endpoints Krickenbeck score, urinary, sexual and QoL evaluation

ELIGIBILITY:
Inclusion Criteria:

Hirschsprung Disease, surgery

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * All Hirschsprung disease patients consecutively
  * Male and female
  * < 18 years
  * Operated by a participating surgeon
  * Elective and emergency surgery
  * Informed consent form signed by the parents of the child
Sampling Method: Non-Probability Sample
Enrollment: 432 (Estimated)
Dates: Start 2012-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To register pre-, intra- and postoperative data in order to improve surgical care to pediatric patients with Hirschsprung's disease in Belgium. | at least 10 years postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium